CLINICAL TRIAL: NCT05534100
Title: Using Wearable Technology to Detect Symptoms of Posttraumatic Stress Disorder
Status: Terminated | Type: Observational
Why Stopped: Trial discontinued due to unreliable wearable device.
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Philip Held, Research Director, Rush University Medical Center
Other Study IDs: 21090706
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control
  Interventions: Device: Biostrap EVO Wristband
- PTSD
  Interventions: Device: Biostrap EVO Wristband

INTERVENTIONS:
Device: Biostrap EVO Wristband — Participants in both groups will wear the Biostrap wearable device

SUMMARY:
The aim of the project is to advance our understanding of how individuals with Posttraumatic Stress Disorder (PTSD) experience symptoms in their every-day lives when they are in their home environment. To date, all PTSD assessments are retrospective; individuals with PTSD are asked to recount and report their symptoms over the past weeks or months. Such assessment procedures are negatively impacted by individuals' abilities to accurately recall information. Moreover, retrospective assessments provide little information about how symptoms are experienced in the moment and how these experiences then lead to other behaviors. The proposed project addresses these limitations by assessing PTSD symptoms and associated biological markers (e.g., sleep, heart rate, heart rate variability) in real-time by asking subjects to wear a smart device and complete brief surveys. Data will be collected from 50 individuals with PTSD and 20 healthy controls to help us better understand individuals' real-time experience with PTSD and lay the foundation to develop algorithms for possible in-the-moment interventions in the future.

ELIGIBILITY:
Inclusion Criteria for participants with PTSD: Individuals are eligible for the current study if they:

1. Are 18 years or older
2. Are fluent in English
3. Have an active smart phone or smart device with full data and Bluetooth capability
4. Have experienced a Criterion A traumatic event during their lifetime
5. Have a PTSD diagnosis verified by the Clinician Administered PTSD Scale for DSM-5 and a symptom severity score of 35 or higher.
6. Are willing and able to complete self-report measures and clinician-rated assessments at multiple time points over the course of the study
7. Are willing to wear a smart device 24/7 over the course of one month.

Exclusion Criteria for PTSD participants: Individuals are excluded from the current study if:

1. The traumatic event occurred in the past month
2. They are currently suicidal or homicidal
3. They have a history of psychosis or mania
4. They have a known, diagnosed heart condition
5. They are currently receiving treatment for their PTSD or have completed an evidence- based PTSD treatment in the past 3 months
6. They have a serious or unstable medical illness or instability for which hospitalization may be likely
7. Subjects who, at the time of consent, appear to have extenuating life circumstances (unstable housing, no internet access, etc.) which, in the judgement of the Principal Investigator, could affect their ability to participate in the study

Inclusion Criteria for healthy controls:

Individuals are eligible for the current study if they:

1. Are 18 years or older
2. Are fluent in English
3. Have an active smart phone or smart device with full data and Bluetooth capability
4. Are willing and able to complete self-report measures and clinician-rated assessments at multiple time points over the course of the study
5. Are willing to wear a smart device 24/7 over the course of one month.

Exclusion Criteria for healthy controls:

Individuals are excluded from the current study if they:

1. Score a 10 or higher on the Clinician Administered PTSD Scale for DSM-5
2. Known or diagnosed heart condition
3. Known or diagnosed psychiatric condition
4. Currently or have previously received psychiatric care in the past 3 months
5. Subjects who, at the time of consent, appear to have extenuating life circumstances (unstable housing, no internet access, etc.) which, in the judgement of the Principal Investigator, could affect their ability to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who either present as a healthy control or are deemed to have PTSD by the CAPS
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale for DSM-5 | Through study completion, average of 1 month
  Clinician administered measure of PTSD
PTSD Checklist for DSM-5 Criteria | Through study completion, average of 1 month
  Self-report measure of PTSD

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No